CLINICAL TRIAL: NCT03445494
Title: Shoulder Abduction Brace Against Normal Sling After Arthroscopical Rotator Cuff Suture: a Randomized Monocentric Study
Brief Title: Shoulder Abduction Brace Against Normal Sling After Arthroscopical Rotator Cuff Suture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Candrian (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, Deputy Head of Surgery and Orthopedy, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-ORT-002
Record Dates: First submitted 2018-01-22; First posted 2018-02-26 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Supraspinatus Injury
MeSH Terms: interventions — Braces

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brace (Experimental): After surgery the patient must wear the brace for 6 weeks, for the first 3 weeks during day and night and for the following 3 weeks only at night
  Interventions: Procedure: Brace
- Normal sling (Experimental): After surgery the patient must wear the normal sling for two weeks
  Interventions: Procedure: Normal sling

INTERVENTIONS:
Procedure: Brace — A brace to be weared according to protocol
  Arms: Brace
Procedure: Normal sling — A normal sling to be weared according to protocol
  Arms: Normal sling

SUMMARY:
The patient undergoes arthroscopic surgery to treat rotator cuff injury. At the end of the surgery, the patient will be randomized into group A (brace) or group B (normal sling).

Both groups will be also treated according to standard of care with physiotherapy and progressive introduction of movements.

DETAILED DESCRIPTION:
The patient undergoes arthroscopic surgery to treat rotator cuff injury. At the end of the surgery, the patient will be randomized into group A (brace) or group B (normal sling).

Both groups will then perform only passive movements according to pain for the first 6 weeks supported by the physiotherapy, according to standard therapy. The following six weeks passive movements will be associated with active movements . No brace nor normal sling will be used anymore.

Patients are in study for 6 months. During this period quality of life and pain questionnaires are submitted to the patients and a MRI will be done at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 65 years old;
* Presence of an isolated lesion of supraspinatus that can be documented with the MRI and which can be treated surgically by arthroscopy;
* Presence of a supraspinatus lesion according to the Patte criteria with stage 1, 2 or 3 frontal plane ;
* Presence of adipose degeneration ≤ 2 according to Goutallier;
* Written informed consent to participate in the study

Exclusion Criteria:

* Presence of a lesion of other rotator cuff tendons;
* Previous surgical procedures of the shoulder;
* Presence of a massive lesion, therefore irreparable, of the cuff detected intra-operatively and not observed during preoperative MRI;
* Presence of relapsing shoulder dislocations;
* Presence of lesions of the glenoidine cercine that require intervention;
* Difficulties to follow the rehabilitation programs;
* Presence of neoplastic diseases, metabolic diseases, inflammatory and systemic diseases, autoimmune diseases and immunosuppressed patients;
* State of pregnancy (presumed or established) or breastfeeding.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Efficacy in the rehabilitative therapy | 6 months
  The primary objective of the study is to evaluate two different rehabilitative therapies. Efficacy is measured with a pre and post MRI

SECONDARY OUTCOMES:
Quality of life assessment | 6 months
  Evaluation of the quality of live in both groups through Constant Quality of Life questionnair up to 6 months
re-rupture rate of the supraspinatus tendon | 6 months
  Evaluation of the re-rupture of the supraspinatus tendon though a follow up MRI at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, MD, Study Director — EOC
Locations (1):
- Ente Ospedaliero Cantonale, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided